CLINICAL TRIAL: NCT01789359
Title: Urinary Excretion of Anthocyanins During Long Term Blueberry Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Food and Horticulture Research Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BBAnthoUrine; AAFC-WBANA (Other Grant/Funding Number: Agriculture & Agri-Food Canada)
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2012-10

CONDITIONS: Bioavailability
Keywords: anthocyanin; bioavailability; urine; long-term

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- anthocyanin-free diet (Other): Maintain anthocyanin-free diet throughout study. Day 1 to day 30, consume daily 250 ml single strength blueberry juice containing 229 mg anthocyanins, taken either as 1 morning dose or 1/3 dose morning, 1/3 mid-day and 1/3 evening. At d 31-38 continue anthocyanin-free diet. On d 39 consume daily dose.
  Interventions: Other: Blueberry Juice

INTERVENTIONS:
Other: Blueberry Juice — Dietary intervention
  Other Names: Single strength wild blueberry juice, commercially prepared.

SUMMARY:
Essentially all of the published data on anthocyanin absorption in humans are from short term studies - a few days or less, most typically 24 h. However human studies demonstrating clinical effects are typically conducted for several weeks or even months. To examine how anthocyanin absorption and metabolism may be affected this study will examine urinary excretion of anthocyanins over one month, followed by a one week washout, and then one more dose of blueberry juice.

ELIGIBILITY:
Inclusion Criteria:

* Provided written consent (see: Information and Consent Form)
* Fluent in English
* Complete a confidential medical questionnaire (Appendix 6)
* Able and willing to abide by the dietary restrictions as described
* Able and willing to abide by the urine collection protocols as described

Exclusion Criteria:

* No written consent
* No confidential medical questionnaire
* Unable to comply with diet restrictions and other study requirements

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Anthocyanins and Phase 2 anthocyanin conjugates in urine | 5 weeks

SECONDARY OUTCOMES:
White blood cell gene expression at start and end of study | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelmina - Kalt, Ph.D., Principal Investigator — Research Scientist
Locations (1):
- Atlantic Food & Horticulture Research Centre, Kentville, Nova Scotia, Canada

REFERENCES:
- [Derived] Kalt W, Liu Y, McDonald JE, Vinqvist-Tymchuk MR, Fillmore SA. Anthocyanin metabolites are abundant and persistent in human urine. J Agric Food Chem. 2014 May 7;62(18):3926-34. doi: 10.1021/jf500107j. Epub 2014 Jan 27. PMID 24432743